CLINICAL TRIAL: NCT01620346
Title: Intracytoplasmic Morphologically Selected Sperm Injection (IMSI) Benefits in the Presence of Advanced Maternal Age: a Prospective Randomized Study
Brief Title: Intracytoplasmic Morphologically Selected Sperm Injection and Advanced Maternal Age
Acronym: IMSIAMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sapientiae Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sapi2012_1
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Female Infertility
Keywords: advanced maternal age; infertility; IMSI; ICSI; implantation
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICSI group (Active Comparator): This group was provided with conventional intracytoplasmic sperm injection (ICSI). This treatment is routinely used to treat infertility. Sperm selection in the ICSI group is analysed under a magnification of 400x using an inverted microscope.
  Interventions: Procedure: Intracytoplasmic sperm injection (ICSI)
- Intracytoplasmic morphologically selected sperm injection (Experimental): Intracytoplasmic morphologically selected sperm injection (IMSI) is an established modified ICSI procedure. Sperm selection in the IMSI group is examined at high magnification using an inverted microscope equipped with high-power differential interference contrast optics (DIC/Nomarski). The total calculated magnification is x6.600. The sperm cells exhibiting normally shaped nuclei and normal nuclear chromatin content are selected for injection.
  Interventions: Procedure: Intracytoplasmic morphologically selected sperm injection

INTERVENTIONS:
Procedure: Intracytoplasmic sperm injection (ICSI) — ICSI is routinely used to treat couples with infertility. Sperm selection in the ICSI group was analysed under a magnification of 400x using an inverted microscope. ICSI was performed in a micro-injection dish prepared with 4 µL droplets of buffered medium (Global® w/HEPES, LifeGlobal, Connecticut, USA) and covered with paraffin oil on a heated stage at 37.0 ± 0.5°C of an inverted microscope.
  Arms: ICSI group
Procedure: Intracytoplasmic morphologically selected sperm injection — IMSI is an established modified ICSI procedure that used an unstained real-time observation of spermatozoa under high-magnification. Sperm selection in the IMSI group is examined at high magnification using an inverted microscope equipped with high-power differential interference contrast optics (DIC/Nomarski). The total calculated magnification is x6.600. The sperm cells exhibiting normally shaped nuclei and normal nuclear chromatin content are selected for injection.
  Arms: Intracytoplasmic morphologically selected sperm injection

SUMMARY:
The objective of this study was to evaluate the advanced maternal age as a rationale for performing intracytoplasmic morphologically selected sperm injection (IMSI).

This prospective randomized study included couples undergoing intracytoplasmic sperm injection (ICSI) as a result of advanced maternal age (≥ 37 years old). Couples were randomly allocated to receive one of two sperm selection procedures (ICSI, n = 33; or IMSI, n = 33). The groups were compared with regard to fertilization rate, percentage of high-quality embryos, implantation, pregnancy and miscarriage rates.

ELIGIBILITY:
Inclusion Criteria:

* Good physical and mental health
* Advanced maternal age (≥ 37 years old)
* Regular menstrual cycles of 25-35 days
* Normal basal FSH and LH levels
* Body mass index less than 30 kg/m2
* Presence of both ovaries
* Intact uterus
* No hormone therapy for at least 60 days preceding the study

Exclusion Criteria:

* Polycystic ovaries
* Endometriosis
* Gynaecological/medical disorders
* Positive result in a screening for sexually transmitted diseases

Min Age: 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 6 weeks after embryo transfer
  Number of embryos implanted in the uterus divided for the number of embryos transferred.

CONTACTS AND LOCATIONS:
Overall Officials: Edson Borges Jr., MD., Ph.D, Principal Investigator — Fertility - Assisted Fertilization Center and Sapientiae Institute - Educational and Research Center in Assisted Reproduction
Locations (1):
- Fertility - Assisted Fertilization Center, São Paulo, São Paulo, Brazil